CLINICAL TRIAL: NCT01564407
Title: A Phase I/II Clinical Study of Allogeneic Human Dermal Fibroblasts for Remodeling Scar Contractures
Brief Title: A Clinical Study of Allogeneic Human Dermal Fibroblasts for Remodeling Scar Contractures
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study Terminated due to lack of Funding
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Prinicipal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO10110342
Record Dates: First submitted 2011-12-20; First posted 2012-03-27 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Restrictive Scar Contracture; Restrictive Hypertrophic Scar; Burn Scar Contractures; Burn Scar
Keywords: ICX-RHY-013; Restrictive scar contracture; Restrictive hypertrophic scar; Burn Scar; Burn Scar contractures; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Safety Cohort (Experimental): Stable restrictive scar contractures resulting from abdominal surgical incision, not transversing a joint. The minimum scar length of 7 cm and a maximum scar area size of 80cm². The scar is divided into five injection areas with a minimum of 0.5 cm uninjected areas between the 5 sites.Drug Dosing for Cohort 1:
  1. Empty control no injection
  2. Vehicle only (0.5 ml of HypoThermosol solution)
  3. 5 million cells / cm² , single administration at Day 0
  4. 5 million cells/ cm² , single administration at week 4
  5. 5 million cells/cm² , single administration at Day 0 , repeat administration of this dose @ week 4 Subjects in Cohort 1 will undergo elective surgeries, at which time the treated scars will be removed, at week 6-8 post-treatment of the first dosed subject.
  Interventions: Drug: ICX-RHY-013
- 2.5M cells/cm2 (Active Comparator): Participants receive intervention treatment of 2.5 million cells/ cm2, single administration injected into the scar.
  Interventions: Drug: ICX-RHY-013
- 5M cells/cm2 (Active Comparator): Participants receive intervention treatment of 5 million cells /cm2, single administration
  Interventions: Drug: ICX-RHY-013
- 2.5M cells/cm2 at 4 weeks (Active Comparator): Participants receive intervention treatment of 2.5 million cells/ cm2, repeat dose administration @ 4 weeks
  Interventions: Drug: ICX-RHY-013
- 5M cells/cm2 at 4 weeks (Active Comparator): Participants receive intervention treatment of 5 million cells / cm2 repeat dose administration @ 4 weeks
  Interventions: Drug: ICX-RHY-013

INTERVENTIONS:
Drug: ICX-RHY-013 — Drug Dosing for Cohorts as follows:
  Cohorts (N=4)
  Safety Cohort 1:
  1. Empty control no injection
  2. Vehicle only (0.5 ml of HypoThermosol solution)
  3. 5 million cells / cm² , single administration at Day 0
  4. 5 million cells/ cm² , single administration at week 4
  5. 5 million cells/cm² , single administration at Day 0 , repeat administration of this dose @ week 4
  At day 0, the subject will receive a total of 3 different injections and at week 4 the subject will receive a total of 2 different injections.
  Cohort 2: 2.5 million cells/ cm2, single administration Cohort 3: 5 million cells /cm2, single administration Cohort 4: 2.5 million cells/ cm2, repeat dose administration @ 4 weeks Cohort 5: 5million cells / cm2 repeat dose administration @ 4 weeks
  Other Names: Allogeneic human dermal fibroblasts

SUMMARY:
The primary objective of this study is to evaluate the safety of ICX-RHY-013 in the treatment of stable, restrictive scars in subjects who have suffered a burn injury. Evaluation will be achieved through regular assessment of adverse events, vital signs, blood work monitoring and laboratory analysis cellular properties of the scar through biopsy.

The secondary objectives of this study are to evaluate improvement in symptoms of scars including reduced pain, discomfort and itching, improvement in mobility and daily function, improvement in appearance and scar texture.

DETAILED DESCRIPTION:
Restrictive scar contracture (a condition where tissue thickens and tightens, pulling the surrounding healthy skin toward the damaged area) due to a serious burn injury can result in long term aesthetic and physical consequences.

Skin contractures adjacent to a joint lead to joint deformities that severely restrict range of motion (ROM) of the affected joint. Skin contractures are also often accompanied by crippling levels of chronic pain resulting in a high level of dependency on pain medications. These isolated or combined factors can lead to a significant disruption in both social and professional life, leading to a marked impact on an individual's quality of life.

The current standard of care for restrictive scar contracture involves the surgical excision of the contracture itself and/ or skin grafting. These standard therapies require extensive and often repeated surgeries. Physicians are continually seeking less invasive therapies to treat patients with burn contractures.

ICX-RHY-013 is an investigational medicinal product comprised of viable allogeneic human dermal fibroblast (HDFs) cells suspended in HypoThermosol®-FRS. HDFs are isolated from neonatal foreskin, cryopreserved, thawed and expanded in culture under good manufacturing practice at Intercytex Ltd., United Kingdom. The drug formulation will be 20 million cells per 1 milliliter of HypoThermosol® and will be administered to subjects via intradermal injections at a maximum dose of 0.25 ml (or 5 million cells) per cm² of tissue.

If determined to be safe and effective, it is believed this therapy could, in the future, be delivered in a series of superficial injections and can be carried out in a doctor's office. This treatment could represent a new less invasive therapy of choice for patients with burn contractures, where current recourse would be to surgery. This advance could have significant positive benefits to the patient in terms of:

* no side-effects of surgery
* treatment given in an outpatient environment without the need for expensive hospitalization
* enhanced quality of life
* lower costs

Cohort 1 will consist of 4 participants who are scheduled to have elective body contouring surgery which will consist of the removal of an abdominal incision scar. The investigational drug will be injected into the existing surgical incision (scar) with the investigational drug, ICX-RHY-013. The purpose of this cohort is to evaluate the initial safety of the investigational drug (ICX-RHY-013) in a series of doses on your surgical scar that will then be surgically removed.

Cohorts 2 through 5 will consist of 4 participants each who have burn scars with restrictive scar contractures. The purpose of these cohorts is to evaluate the ongoing safety of the investigational drug (ICX-RHY-013) in post burn scars with restrictive scar contractures. The investigational drug will be injected directly into these scar contractures. Each cohort is unique in that the dose and frequency of the investigational drug received will be different. We will evaluate the safety of the drug between each cohort by assessing all side effects that the participants may experience.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are male or female, military or civilian, age 18 to 65 years of age and able to provide informed consent
2. Subjects who have suffered an injury which has occurred no less than 6 weeks prior to their screening date which has resulted in a stable restrictive scar contracture

   1. Stable restrictive scar contracture that has resulted from abdominal surgical incision and does not transverse a joint (Cohort 1 only).
   2. Stable restrictive scar contracture has resulted from a burn injury and may transverse a joint (Cohorts 2-5 only)
3. Subjects will have a minimum scar length of 7 cm and a maximum scar area size of 80cm² (Cohort 1 only)
4. Subjects will have a minimum scar area size of 1cm² and a maximum scar area size of 80cm² (Cohort 2-5 only).
5. Subjects who are, in the opinion of the Investigator, able to understand the study, comply with the study design and are willing to return to the clinic for all the research required follow-up visits

Exclusion Criteria:

1. Subjects with previous use of cellular therapy (e.g. Isolagen) in the treatment area
2. Subjects with a known history of keloids
3. Subjects with a known history of bleeding disorders
4. Subjects who have facial restrictive scar deficits, not to exclude the neck area.
5. Subjects who have had contracture-release procedures in the treatment area within the previous six months
6. Subjects with a known allergy to any of the constituents of HypoThermosol-FRS
7. Subjects taking immunosuppressive therapy including systemic steroids will be excluded if they have received any dose >7.5 mg of prednisone equivalent/day for more than one week within 90 days of the first treatment or planning immunosuppressive therapy at any time during the study (Intranasal/inhaled steroids are acceptable)
8. Diagnosis of cancer within last 12 months and /or actively receiving chemotherapy or radiation treatment
9. Subjects with a life expectancy of <9 months, terminal conditions or factors making follow-up difficult (e.g. no fixed address, telephone etc)
10. Subjects with a history of hypersensitivity to additional study-associated drugs/therapies (e.g. isopropyl alcohol, EMLA cream, adrenaline, lidocaine, etc)
11. Subjects with planned major surgical intervention during the course of the study.
12. Subjects with known idiopathic or drug-associated coagulopathy
13. Subjects taking medicinal products known to reduce hemostasis (e.g. heparin, Coumadin, etc.) in the 2 weeks prior to commencing treatment or planning to take medicinal products known to reduce hemostasis during the 12 week study period
14. Subjects who have taken any other investigational product within 30 days prior to screening or planned use of any other investigational product during the study period.
15. Subjects who are pregnant, lactating, planning pregnancy and women of child-bearing potential who are not abstinent or practicing an acceptable means of contraception, as determined by the Investigator, for the duration of the treatment phase
16. Subjects with abnormal blood biochemistry or any other abnormal laboratory finding considered clinically significant in that it would deem the subject inappropriate for surgical procedures, as determined by the investigator (i.e. CBC with Differential, platelets, comprehensive metabolic panel to include electrolytes, bun/creatinine, liver function test and coagulation tests).
17. Subjects who have, as determined by the investigator a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study (i.e. Type 1 and Type 2 diabetic patients) or any condition within the last 14 days requiring hospitalization or surgical intervention.
18. Subjects with evidence of any past or present clinically significant medical condition that would impair wound healing
19. Subjects with a known hypersensitivity to gentamycin, amphotericin B, Bovine serum or porcine products.
20. Subjects with known alcohol or narcotic drug dependency
21. Subjects with diagnosed autoimmune disorders known to affect wound healing, such as Systemic Lupus Erythematosis (SLE), psoriasis, infection and inflammation (seborrheic dermatitis).
22. Subjects receiving an immunosuppressive medication regime including transplant anti-rejection agents.
23. Subjects with an Axis II to diagnosis DSM-IV (e.g., Schizophrenia, Bipolar Disorder). Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multiple approaches for subject recruitment were implemented.The Center for Innovation in Restorative (CIRM) hired a marketing specialist who investigated the use of non-traditional mechanisms within and outside the existing infrastructure including but not limited to social media outlet,use of internal/external physician networks,TV advertising
Pre-assignment Details: All of the subjects who were enrolled (signed consent) were randomized to 1 of 4 cohorts.
Groups:
- No Injection: Safety cohort. 4 subjects received empty control. No injection
- Vehicle Only: Vehicle only (0.5 ml of solution)
- Single Admin Drug Day 0: Single administration of study drug on day 0
- Single Admin Drug Day 28: Single administration on Day 28
- Admin Drug Day 0 and 28: Single administration day 0 and 28
Period: Overall Study
Arm/Group | No Injection | Vehicle Only | Single Admin Drug Day 0 | Single Admin Drug Day 28 | Admin Drug Day 0 and 28
Started | 4 | 5 | 4 | 2 | 0
Completed | 4 | 3 | 4 | 1 | 0
Not Completed | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — funding lost, study ended | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Injection: Empty safety control, no injection
- Vehicle Only: Vehicle only (0.5 ml of HypoThermosol solution)
- Single Admin Day 0: 5 million cells / cm² , single administration at Day 0
- Single Admin Day 28: 5 million cells/ cm² , single administration at day 28
- Admin Day 0 and 28: 5 million cells/cm² , single administration at Day 0 , repeat administration of this dose @ day 28
- Total: Total of all reporting groups
Arm/Group | No Injection | Vehicle Only | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 0 | 15
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 4 | 5 | 4 | 2 |  | 15
  >=65 years | 0 | 0 | 0 | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.25 (12.3) | 41.25 (17.0) | 45.75 (14.9) | 62 (0) |  | 45.3 (12.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 4 | 1 | 0 | 0 |  | 5
  Male | 0 | 4 | 4 | 2 |  | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 2 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The evaluation of safety of ICX-RHY-013 in the treatment of stable, restrictive hypertrophic scars through assessment of adverse events. The primary objective of the safety (no injection) cohort is to evaluate initial safety of multiple doses through assessment of adverse events. The primary objective of remaining cohorts is to evaluate the ongoing safety of ICX-RHY-013 in post-burn hypertrophic scars that are not planned for excision through assessment of adverse events.
Time Frame: Days 0, 7, 14, 28, 56, 84
Measure: Number; unit: participants
Groups:
- no Injection: Empty control no injection
- Single Admin Drug Day 28: Single administration of study drug on day 28
Arm/Group | no Injection | Vehicle Only | Single Admin Drug Day 0 | Single Admin Drug Day 28
Number analyzed (Participants) | 4 | 3 | 4 | 1
participants | 4 | 3 | 4 | 1

2. Primary Outcome: Number of Participants With Serious Adverse Events Reported
Description: The evaluation of tolerability of ICX-RHY-013 in the treatment of stable, restrictive hypertrophic scars through regular assessment of adverse events.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | No Injection | Vehicle Only | Single Admin Drug Day 0 | Single Admin Drug Day 28
Number analyzed (Participants) | 4 | 3 | 4 | 1
participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Subjects Worse Hypertrophic Scars
Description: The secondary objectives of this study are to evaluate improvement in symptoms of hypertrophic scars.
Time Frame: Endpoints assessed at Day 84.
Measure: Number; unit: percentage of paricipants
Arm/Group | no Injection | Vehicle Only | Single Admin Drug Day 0 | Single Admin Drug Day 28
Number analyzed (Participants) | 4 | 3 | 4 | 1
percentage of paricipants | 0 | 0 | 0 | 0

4. Secondary Outcome: Vancouver Scar Scale
Description: Vancouver scar scale will be evaluated for each cohort. The Vancouver scar scale is the most frequently cited assessment of scar severity used in clinical studies. Pigmentation, vascularity, pliability, and scar height are graded producing a composite score. A score of 0 represents normal skin with higher grades representing greater deformity with a maximum possible rating of 14.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | No Injection | Vehicle Only
Number analyzed (Participants) | 4 | 2 | 0 | 4 | 5
scores on a scale | 8 (2) | 10 (2.2) |  | 10 (3) | 8 (1.3)

5. Secondary Outcome: Patient and Observer Scar Assessment Scale (POSAS)
Description: POSAS aims to measure scar quality, it is a comprehensive scale designed for the evaluation of all types of scars by professionals and patients. It contains two scales with six items, scored numerically from 0-10, where 0 is normal skin and 10 is the worst scar imaginable. the total scoring range is from 0-120.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | No Injection | Vehicle Only
Number analyzed (Participants) | 4 | 2 | 0 | 4 | 5
scores on a scale | 24.67 (1.53) | 34.25 (11.32) |  | 42.13 (8.16) | 41.57 (4.32)

6. Secondary Outcome: Disability Index-Disability of Arm, Shoulder and Hand
Description: The six subjects suffering from upper extremity and cervical scar contractures were evaluated with the Disability of Arm, Shoulder and Hand (DASH) questionnaire. The DASH questionnaire evaluates symptoms and functional status. A lowest score of 0 indicates normal skin and highest score of 100 represents the greatest possible morbidity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | No Injection | Vehicle Only
Number analyzed (Participants) | 4 | 2 | 0 | 4 | 5
scores on a scale | 6.9 (6) | 11.6 (14.1) |  | 75.5 (3.8) | 69.2 (12.7)

7. Secondary Outcome: Quality of Life Measurement - Satisfaction With Appearance Scale (SWAP)
Description: SWAP is a psychological test for personality diagnosis. there are 9 questions evaluated by a score of 7 (most descriptive to the patient) to 0 (not descriptive or irrelevant) for a total scoring range of 0-63.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | No Injection | Vehicle Only
Number analyzed (Participants) | 4 | 2 | 0 | 4 | 5
units on a scale | 5.67 (7.37) | 37.75 (14.73) |  | 13.35 (4.12) | 23.27 (9.87)

ADVERSE EVENTS:
Groups:
- Vehicle Only,; Single Admin Day 0; Single Admin Day 28; Admin Day 0 and 28; no Injection: Adverse events in each cohort included pain, swelling and redness at the site of injection that resolved within 8 hours of treatment
Arm/Group | Vehicle Only, | Single Admin Day 0 | Single Admin Day 28 | Admin Day 0 and 28 | no Injection
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/2 | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/2 | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 2/2 | 0/0 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Only, (N=5) | Single Admin Day 0 (N=4) | Single Admin Day 28 (N=2) | Admin Day 0 and 28 (N=0) | no Injection (N=4)
Redness (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Warmth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Bleeding from injection and also biopsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No